CLINICAL TRIAL: NCT02400320
Title: Cumulative Skin Irritation Study Evaluating the Skin Irritancy Potential of Topical Analgesic Vovilup Spray Containing a Combination of Diclofenac, Menthol, Methyl Salicylate and Linseed Oil and Comparing it With a Marketed Formulation - Iodex Ultragel
Brief Title: Local Skin Safety Study of a Topical Pain Relief Spray Containing a Combination of Diclofenac, Methyl Salicylate, and Menthol
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202201
Record Dates: First submitted 2015-01-29; First posted 2015-03-27 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Skin Irritation
MeSH Terms: interventions — Gels; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Topical Spray (Active Comparator): Topical spray containing Diclofenac 1.16%, Linseed Oil 3%, Menthol 5%, Methyl salicylate 10%.
  Interventions: Drug: Topical Spray
- Topical Gel (Experimental): Topical gel containing Diclofenac 1.16%, Menthol 5%, Methyl salicylate 10%
  Interventions: Drug: Topical Gel
- Saline (Other): Saline
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Topical Spray — Topical spray containing Diclofenac 1.16%, Linseed Oil 3%, Menthol 5%, Methyl salicylate 10%.
  Arms: Topical Spray
Drug: Topical Gel — Topical gel containing Diclofenac 1.16%, Menthol 5%, Methyl salicylate 10%
  Arms: Topical Gel
Other: Saline — Saline
  Arms: Saline

SUMMARY:
The purpose of this study is to determine local skin safety of a topical analgesic spray containing a combination of diclofenac, methyl salicylate, menthol and compare it with a topical analgesic gel containing a combination of diclofenac, methyl salicylate, and menthol.

ELIGIBILITY:
Inclusion Criteria

1. Healthy male or female volunteers aged at least 18 years.
2. Good general, physical and mental health in the opinion of the investigator or medically qualified designee:

   * No clinically significant and relevant abnormalities in medical history or upon physical examination.
   * Absence of any condition that could affect the volunteer's safety or well being or their ability to understand and follow study procedures and requirements.
3. Healthy volunteers who do not have excessive hair on the volar aspect of the forearm(s).
4. Healthy volunteers should understand and be willing to fully comply with all study procedures and restrictions.
5. Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
6. Females of childbearing potential, using an effective contraceptive method for at least one month before the beginning of the study, and willing to use throughout the study

Exclusion Criteria

1. Volunteers having recent history (within one year) of alcohol or other substance abuse as determined by medical history.
2. Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
3. Previous participation in similar study with similar products.
4. Volunteer has any visible skin disease at the site of application that, in the opinion of the investigator, will interfere with the skin assessments.
5. Volunteer has current or relevant previous history of serious, severe or unstable physical or psychiatric illness, or medical disorders, such as current or previous history of hepatic or renal diseases (impairment) or peptic ulcer as determined by medical history.
6. Volunteer has a history of hypersensitivity (e.g. asthma, bronchospasm, rhinitis, urticaria, nasal polyps) to aspirin, diclofenac, other non steroidal anti-inflammatory drugs (NSAIDs), menthol or any of the excipients in the test product(s).
7. Volunteer is receiving systemic or topical NSAIDs, other oral or topical analgesics or antihistamine within 3 days of visit 1, or other medication (such as corticosteroids within 3 weeks of visit 1) which, in the opinion of the investigative personnel, will interfere with the study results.
8. Female volunteers who are pregnant, planning to become pregnant during the study, or are breast-feeding.
9. Female volunteers who have positive pregnancy test.
10. Volunteers who are employees of the sponsor or study site or an immediate family member (e.g. partner, offspring, parents, siblings or sibling's offspring) of such employees.
11. Any skin disorder at the test site that in the investigator's judgement can affect the readings of the test result
12. Any concomitant medications that in the investigator's judgement can confound or alter test results or evaluation of adverse events.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-01 (Estimated); Primary Completion 2016-06-01 (Estimated); Study Completion 2016-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean cumulative irritation score | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline